CLINICAL TRIAL: NCT00270764
Title: Economic Outcomes of HIV/AIDS Care and Treatment in South Africa
Brief Title: Social and Economic Outcomes of HIV/AIDS Care and Treatment in HIV Infected South African Adults
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: PEPFAR 13
Record Dates: First submitted 2005-12-27; First posted 2005-12-28 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections
Keywords: HIV/AIDS; Antiretroviral therapy; Quality of life; South Africa; Treatment Naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Full cohort: Adult ART patients at 3 treatment facilities in South Africa

SUMMARY:
The purpose of this study is to determine the social and economic outcomes of anti-HIV treatment in South African adults, with data collected from interviews, detailed questionnaires, and patients' medical records.

DETAILED DESCRIPTION:
The Government of the Republic of South Africa is implementing a national program to provide antiretroviral therapy (ART) to all eligible HIV infected South African adults. While the medical effectiveness of ART in suppressing viral replication is well established, little is known about the economic effectiveness of treatment. In particular, it is not known if treatment will offset the impact of HIV/AIDS on labor productivity, household stability, quality of life, and other aspects of social and economic development. The purpose of this study is to estimate the impact of ART on the productivity, economic welfare, and quality of life of adult HIV infected patients in South Africa. The study will investigate:

* the degree of functional impairment among patients seeking care for HIV/AIDS,
* the impact of treatment on the ability of patients to perform normal daily activities and attend work,
* the full economic costs to patients of obtaining treatment,
* the impact of treatment on sources of household income,
* social and economic correlates of adherence to therapy, and
* the cost of delivering ART to different types of patients in diverse settings.

The study will last 4 years and will comprise a one-year cross-sectional analysis and a three-year longitudinal analysis. Data will be collected from questionnaires administered during patients' routine visits to public and non-governmental organization-based HIV clinics in South Africa. In accordance with current South African national treatment guidelines, patients who have started ART will visit a clinic every 3 months during the longitudinal analysis for a total of 12 visits; patients not yet on ART will visit a clinic every 6 months for a total of 6 visits.

Questionnaire responses will be matched to indicators of disease progression and treatment history drawn from patients' medical records. The initial one-year analysis will compare outcomes for groups of patients stratified by disease stage and treatment duration. Longitudinal analysis will compare outcomes before and after the initiation of ART; each participant's responses and medical outcomes will be compared with his or her own previous results and with those of other participants at a similar stage of disease progression or treatment duration. This study will generate information needed to sustain large-scale treatment interventions, improve the focus and management of treatment delivery programs, and provide a better understanding of barriers to treatment adherence among HIV infected South African patients.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Willing to accept ART if medically eligible according to South Africa's national treatment guidelines

Exclusion Criteria:

* Inability to answer questions due to disability
* On ART for more than 6 months at the time of study entry
* Refuse to accept ART despite medical eligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ART patients receiving treatment at 3 treatment facilities in South Africa
Sampling Method: Probability Sample
Enrollment: 1065 (Actual)
Dates: Start 2005-07; Primary Completion 2011-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Ability to perform normal activities in previous week | Previous week

CONTACTS AND LOCATIONS:
Overall Officials: Sydney B. Rosen, MPA, Principal Investigator — Boston University
Locations (1):
- Health Economics Research Office, Helen Joseph Hospital, Johannesburg, Gauteng, South Africa

REFERENCES:
- [Background] Beard J, Feeley F, Rosen S. Economic and quality of life outcomes of antiretroviral therapy for HIV/AIDS in developing countries: a systematic literature review. AIDS Care. 2009 Nov;21(11):1343-56. doi: 10.1080/09540120902889926. PMID 20024710
- [Result] Rosen S, Ketlhapile M, Sanne I, Desilva MB. Differences in normal activities, job performance and symptom prevalence between patients not yet on antiretroviral therapy and patients initiating therapy in South Africa. AIDS. 2008 Jul;22 Suppl 1:S131-9. doi: 10.1097/01.aids.0000327634.92844.91. PMID 18664945
- [Result] Rosen S, Ketlhapile M, Sanne I, DeSilva MB. Characteristics of patients accessing care and treatment for HIV/AIDS at public and nongovernmental sites in South Africa. J Int Assoc Physicians AIDS Care (Chic). 2008 Jul-Aug;7(4):200-7. doi: 10.1177/1545109708320684. Epub 2008 Jul 14. PMID 18626120
- [Result] Rosen S, Ketlhapile M, Sanne I, DeSilva MB. Cost to patients of obtaining treatment for HIV/AIDS in South Africa. S Afr Med J. 2007 Jul;97(7):524-9. PMID 17805455
- [Result] Rosen S, Larson B, Brennan A, Long L, Fox M, Mongwenyana C, Ketlhapile M, Sanne I. Economic outcomes of patients receiving antiretroviral therapy for HIV/AIDS in South Africa are sustained through three years on treatment. PLoS One. 2010 Sep 14;5(9):e12731. doi: 10.1371/journal.pone.0012731. PMID 20856821
- [Result] Rosen S, Larson B, Rohr J, Sanne I, Mongwenyana C, Brennan AT, Galarraga O. Effect of antiretroviral therapy on patients' economic well being: five-year follow-up. AIDS. 2014 Jan 28;28(3):417-24. doi: 10.1097/QAD.0000000000000053. PMID 24076660